CLINICAL TRIAL: NCT03328416
Title: Augmented Reality Headset as Adjunct Display Monitor in AMIGO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Expected technology was not available.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas C. Lee, Assistant Professor of Radiology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P001456
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Malignancy; Infection; Pain
Keywords: Image-Guided Biopsy; Multidetector Computed Tomography; Diagnostic Imaging; Cryosurgery; Ablation Techniques
MeSH Terms: conditions — Neoplasms; Infections; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented Reality (Experimental): The neurointerventional radiologist will have imaging information projected on a headset in addition to on the conventional monitors that hang from the procedure suite ceiling.
  Interventions: Device: Augmented Reality

INTERVENTIONS:
Device: Augmented Reality — The neurointerventional radiologist will have imaging information projected on a headset in addition to on the conventional monitors that hang from the procedure suite ceiling.

SUMMARY:
The investigators' overarching goal is to investigate whether use of an augmented reality display system (utilized in addition to, not as a replacement to, conventional CT and MRI displays currently available in the procedure suite) streamlines the process of a procedure and/or provides ease of access to helpful pre-procedure and intra-procedure imaging information that would be more difficult and time-consuming to obtain with the conventional imaging display systems.

DETAILED DESCRIPTION:
Augmented reality is a computer display technology that represents an incremental improvement over current computer monitors. Currently, a patient has a pre-procedure or intra-procedure CT or MRI scan and the scan images are displayed for the proceduralist on computer monitors in the procedure suite. Typically, only a single, or several selected, cross-sectional images can be viewed at a given time. With an augmented reality display headset, the pre-procedure and intra-procedure CT or MR images, including 3D reconstructions, can be displayed on transparent eyeglasses worn by the proceduralist. Moreover, the images are registered to the patient's location on the operating table and the images can be continuously updated to correspond with the body part in the proceduralist's field of view. Augmented reality display systems could thus decreased perceived work load of a procedure by allowing natural posture throughout the procedure, streamline and improve the clinical workflow, and provide the proceduralist with information in a manner that more readily facilitates three-dimensional understanding of the procedure.

The investigators' overarching goal is to investigate whether use of an augmented reality display system (utilized in addition to, not as a replacement to, conventional CT and MRI displays currently available in the procedure suite) streamlines the process of a procedure and/or provides ease of access to helpful pre-procedure and intra-procedure imaging information that would be more difficult and time-consuming to obtain with the conventional imaging display systems.

The three aims are as follows:

1. Determine if the augmented reality display system streamlines workflow.
2. Determine if the augmented reality display system decreases perceived work load.
3. Determine if the augmented reality display system facilitates access to helpful pre-procedure and intra-procedure imaging information as compared to traditional display systems.

The investigators hypothesize that the augmented reality display system will streamline workflow by reducing time required to stop the procedure to look away from the operative field to the conventional hanging monitor and then look back to the operative field and reorient to the operative field space.

The investigators hypothesize that the augmented reality display system will decrease perceived work load by reducing intra-procedure postural strain by projecting the images on a headset in addition to on traditional monitors hanging from the procedure-suite ceiling.

The investigators hypothesize that the augmented reality display system will facilitate access to helpful pre-procedure and intra-procedure imaging information because it will allow real-time projection of three-dimensional reconstructed images over the operative site with the images reflecting the point-of-view and field-of-view of the proceduralist. While this information can be generated and projected on traditional display systems, the positioning of the imaging is likely inferior as it can only mimic the point of view and field of view of the proceduralist.

All procedures will be performed in accordance with normal standard of care for the condition being treated. The only difference in care will be that the proceduralist will have imaging information projected on a headset in addition to on the conventional monitors that hang from the procedure suite ceiling.

A single REDCap survey will be sent to the performing co-investigator proceduralist (interventional radiologist or surgeon) following each procedure. The survey will include the NASA Task Load Index (TLX) to assess the work load associated with the procedure as well as several questions designed to determine if the NASA TLX score would likely have been higher or lower if the augmented reality system was not used and several questions designed to determine if the augmented reality system allowed visualization of imaging information in a way that was helpful in procedure planning or intraprocedural approach. The NASA TLX method assesses work load on five 7-point scales and the additional questions assess procedural strain on 7-point scales.

The primary outcome measures are the TLX scores. If these scores achieve statistical significance in one sample statistical tests then use of the augmented reality display will be considered successful. Although co-investigators will be subjects, the co-investigators have no relationship with the device maker and have no invested interest in using this device unless the device improves procedure efficiency and success; as such, it is unlikely that co-investigators as subjects will bias the results as the co-investigators will not want to utilize the device if it has a negative impact on workflow or if it increases perceived work load.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred to one of the study co-investigators for a procedure that requires either: Pre-procedure planning that utilizes either CT or MR images; Intra-procedure imaging for the purpose of needle placement.

Exclusion Criteria:

* Age under 18 at time of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Scores from NASA Task Load Index (TLX) with supplemental questions to assess procedure strain | 15 minutes
  The NASA TLX method assesses work load on five 7-point scales and the additional questions assess procedural strain on 7-point scales. Each 7-point scale item will be assessed independently. Total scores will also be summed and assessed. Higher scores translate to a higher work load (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Lee, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided